CLINICAL TRIAL: NCT02122211
Title: Choline Dehydrogenase and Sperm Function: Effects of Betaine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-2424
Record Dates: First submitted 2014-04-17; First posted 2014-04-24 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Men Carrying 2 Minor Alleles for Choline Dehydrogenase rs12676; Male Infertility
Keywords: Sperm motility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Betaine supplement (Experimental): Will use powdered betaine (BetaPower, Dupont Nutrition) that is commercially available for food uses. This powder will be delivered as capsules containing 0.5 gram of powdered betaine which will be administered as eleven capsules twice per day (6 in the morning, 5 in the evening) for a daily total of 6 grams of betaine.
  Interventions: Drug: Betaine supplement

INTERVENTIONS:
Drug: Betaine supplement
  Other Names: BetaPower (Dupont Nutrition)

SUMMARY:
The ability of sperm to swim is important for normal fertility. Men with a genetic variation in the gene coding for Choline Dehydrogenase (CHDH) have decreased energy production by sperm, and their sperm do not swim normally. The metabolic product of this gene is a nutrient called betaine (found normally in the diet as a part of many foods such as spinach, beets and grain products). This study tests whether treatment with betaine is safe and whether it can normalize energy production in sperm of these men and restore normal swimming ability.

DETAILED DESCRIPTION:
Unidentified genetic aberrations such as single nucleotide polymorphisms (SNPs) may be the underlying cause of many cases of idiopathic infertility in men. Choline dehydrogenase (encoded by CHDH) converts choline to betaine in the mitochondria. 5-9% of men have 2 alleles for a functional SNP in CHDH (rs12676), and they have low sperm adenosine triphosphate (ATP) concentrations with impaired sperm motility (asthenospermia) that should decrease fertility. Male mice in which CHDH is deleted also have very low sperm ATP, asthenospermia and are infertile. Supplementation of these mice with dietary betaine increases sperm motility and ATP concentrations.

This purpose of this study is to conduct a phase I study of betaine treatment in men with 2 minor alleles for CHDH rs12676 to determine whether betaine supplementation is safe and to obtain preliminary data on the effects of betaine on sperm mitochondrial ATP concentrations and sperm motility in these men.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 60 year old men of multiple races and ethnicities
* Estimated dietary intake of betaine of <150 mg/day
* Carrying two alleles of the rs 12676 single nucleotide polymorphism

Exclusion Criteria:

* Cystathionine-beta-synthase (CBS) deficiency
* Currently taking betaine supplements
* Currently receiving chemotherapy, radiation or any gonadotoxic drug
* Female gender

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in sperm motility from baseline | On day zero, day 10, day 30, day 50 and at the end of the 75 day treatment period
  Assessed using Computer-Aided Sperm Analysis methodology
Change in sperm count from baseline | On day zero, day 10, day 30, day 50 and at the end of the 75 day treatment period
Change in sperm mitochondrial function from baseline | On day zero, day 10, day 30, day 50 and at the end of the 75 day treatment period
  Using Seahorse biochemical function assessment
Change in sperm ultrastructure from baseline | On day zero, day 10, day 30, day 50 and at the end of the 75 day treatment period
  Using light and transmission electron microscopy
Change in sperm choline dehydrogenase concentration from baseline | On day zero, day 10, day 30, day 50 and at the end of the 75 day treatment period
  Assessed by Western Blot analysis
Change in sperm betaine concentration from baseline | On day zero, day 10, day 30, day 50 and at the end of the 75 day treatment period

SECONDARY OUTCOMES:
Betaine intake | At screening and every 21 days during the study
  Assessed using 3-day food records
Change in complete blood count from baseline | At 0, 10, 30, 50, and 75 days on treatment
Change in uric acid concentration from baseline | At 0, 10, 30, 50, and 75 days on treatment
Change in alkaline phosphatase concentration from baseline | At 0, 10, 30, 50, and 75 days on treatment
Change in aspartate transaminase concentration from baseline | At 0,10, 30, 50, and 75 days on treatment
Change in lactic dehydrogenase concentration from baseline | At 0, 10, 30, 50, and 75 days on treatment
Change in bilirubin concentration from baseline | At 0, 10, 30, 50, and 75 days on treatment
Change in blood urea nitrogen concentration from baseline | At 0, 10, 30, 50, and 75 days on treatment
Change in creatinine concentration from baseline | At 0, 10, 30, 50, and 75 days on treatment
Change in urinalysis parameters from baseline | At 0, 10, 30, 50, and 75 days on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steven Zeisel, MD, PhD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Nutrition Research Institute, Kannapolis, North Carolina, United States

REFERENCES:
- [Background] Johnson AR, Lao S, Wang T, Galanko JA, Zeisel SH. Choline dehydrogenase polymorphism rs12676 is a functional variation and is associated with changes in human sperm cell function. PLoS One. 2012;7(4):e36047. doi: 10.1371/journal.pone.0036047. Epub 2012 Apr 27. PMID 22558321